CLINICAL TRIAL: NCT03731195
Title: GentleTouch (Study to Evaluate Somatosensory Evoked Potential (SSEP) Responses to Affective Touch and How it Develops in Healthy Term Babies)
Status: Completed | Type: Observational
Sponsor: University College Cork (Other)
Collaborators: University College London - Institute of Child Health (UCL-ICH) (Unknown); Science Foundation Ireland (Other); Johnson & Johnson (Industry)
Responsible Party: Principal Investigator, Professor Geraldine Boylan, Professor of Neonatal Physiology and Director of INFANT Centre, University College Cork
Other Study IDs: GB01/18UCC
Record Dates: First submitted 2018-11-02; First posted 2018-11-06 (Actual); Last update posted 2023-12-11 (Actual); Status verified 2023-12

CONDITIONS: Pleasant Touch; Cortical Response
Keywords: Baby Massage; SSEP

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will attempt to measure the direct effect of pleasant skin touch on the developing infant brain. The massage intervention stimulates a specific class of unmyelinated C-fibres in the skin called C-touch (CT) afferents, and effects will be assessed by monitoring brain responses (GentleTouch Project) in a prospective cohort study.

DETAILED DESCRIPTION:
This is a single-centre proof of concept translational study to determine how and when Somato-sensory evoked potentials develop over the first 4 months of life.

The aim of this study is to explore if the investigators can measure the cortical response from the scalp of infants using standard non-invasive EEG techniques, due to the activation of CT afferents and explore how the cortical response changes in regard to age. Preform a longitudinal study on 40 subjects at approximately 4 weeks and 4 months of age. The Gentle Touch study will examine the effect of gentle positive stimuli applied to an infant's forearm on cortical responses at two time points within the first 4 months of life.

ELIGIBILITY:
Inclusion Criteria:

* Infants born > 37 weeks gestation
* Single births
* Not requiring admission to the Neonatal Unit
* Healthy infants without suspected congenital or metabolic anomalies
* Written Informed Consent

Exclusion Criteria:

* Infants born < 37 weeks gestation
* Multiple births
* Severe metabolic or genetic anomaly that would require ongoing specialist care in the infancy period.
* Admission to the Neonatal Unit.
* No written Informed Consent obtained

Min Age: 37 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Healthy Term infants >37 weeks Gestational Age
Sampling Method: Non-Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2020-12-30 (Actual); Study Completion 2021-07-08 (Actual)

PRIMARY OUTCOMES:
Measurement and development of SSEP response to positive touch stimuli | 4 weeks
  Standard Evoked Potentials

SECONDARY OUTCOMES:
Measurement of SSEP to positive touch stimuli | 4 months
  Standard Evoked Potentials
Neurodevelopmental Assessment | 4 months
  Griffiths Mental Development Scales (GMDS)Griffiths III provides an overall measure of a child's development, as well as an individual profile of strengths and needs across five areas:
  * Foundations of Learning
  * Language and Communication
  * Eye and Hand Coordination
  * Personal-Social-Emotional
  * Gross Motor
  Very Superior 16-20 Scaled Score >130 Development Quotient Superior 14- <16 Scaled Score 120 - 129 Development Quotient Above Average 12- <14 Scaled Score 110 - 119 Development Quotient Average 8- <12 Scaled Score 90 - 109 Development Quotient Below Average 6- <8 Scaled Score 80 - 89 Development Quotient Borderline 4- <6 Scaled Score 70 - 79 Development Quotient Extremely Low 0- <4 Scaled Score ≤ 69 Development Quotient

CONTACTS AND LOCATIONS:
Overall Officials: Ronit Pressler, MD, Principal Investigator — University College London - Institute of Child Health (UCL-ICH)
Locations (2):
- Cork University Maternity Hospital, Wilton, Cork, Ireland
- University College London - Institute of Child Health (UCL-ICH), London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Ventura S, Mathieson SR, O'Toole JM, Livingstone V, Ryan MA, Boylan GB. Electroencephalographic sleep macrostructure and sleep spindles in early infancy. Sleep. 2022 Jan 11;45(1):zsab262. doi: 10.1093/sleep/zsab262. PMID 34755881
- [Result] Wei L, Ventura S, Mathieson S, Boylan G, Lowery M, Mooney C. Spindle-AI: Sleep Spindle Number and Duration Estimation in Infant EEG. IEEE Trans Biomed Eng. 2022 Jan;69(1):465-474. doi: 10.1109/TBME.2021.3097815. Epub 2021 Dec 23. PMID 34280088
- [Result] Wei L, Ventura S, Ryan MA, Mathieson S, Boylan GB, Lowery M, Mooney C. Deep-spindle: An automated sleep spindle detection system for analysis of infant sleep spindles. Comput Biol Med. 2022 Nov;150:106096. doi: 10.1016/j.compbiomed.2022.106096. Epub 2022 Sep 15. PMID 36162199
- [Result] Wei L, Ventura S, Lowery M, Ryan MA, Mathieson S, Boylan GB, Mooney C. Random Forest-based Algorithm for Sleep Spindle Detection in Infant EEG. Annu Int Conf IEEE Eng Med Biol Soc. 2020 Jul;2020:58-61. doi: 10.1109/EMBC44109.2020.9176339. PMID 33017930
- [Result] Lenehan SM, Fogarty L, O'Connor C, Mathieson S, Boylan GB. The Architecture of Early Childhood Sleep Over the First Two Years. Matern Child Health J. 2023 Feb;27(2):226-250. doi: 10.1007/s10995-022-03545-9. Epub 2022 Dec 31. PMID 36586054
- [Result] O Sullivan MP, Livingstone V, Korotchikova I, Dempsey EM, Murray DM, Boylan GB. Reference centiles for infant sleep parameters from 4 to 16 weeks of age: findings from an Irish cohort. Arch Dis Child. 2023 Jun;108(6):481-485. doi: 10.1136/archdischild-2022-324016. Epub 2023 Mar 21. PMID 36944485
- [Result] Ventura S, Mathieson SR, O'Sullivan MP, O'Toole JM, Livingstone V, Pressler RM, Dempsey EM, Murray DM, Boylan GB. Parent-led massage and sleep EEG for term-born infants: A randomized controlled parallel-group study. Dev Med Child Neurol. 2023 Oct;65(10):1395-1407. doi: 10.1111/dmcn.15565. Epub 2023 Mar 14. PMID 36917624